CLINICAL TRIAL: NCT02182752
Title: The Effect of Tramadol on Interscalene Brachial Plexus Block With Ropivacaine in Shoulder Surgery.
Brief Title: The Effect of Tramadol on Interscalene Brachial Plexus Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Collaborators: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Eleftheria Soulioti, MD, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3694/27-3-13
Record Dates: First submitted 2014-06-30; First posted 2014-07-08 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Shoulder Fracture; Shoulder Dislocation; Rotator Cuff Injury; Shoulder Arthritis
MeSH Terms: conditions — Shoulder Fractures; Shoulder Dislocation; Rotator Cuff Injuries | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ropivacaine - Tramadol (Active Comparator)
  Interventions: Drug: Ropivacaine - Tramadol
- Ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine - Tramadol — Interscalene block using ropivacaine plus tramadol
  Arms: Ropivacaine - Tramadol
Drug: Ropivacaine — Interscalene block using ropivacaine
  Arms: Ropivacaine

SUMMARY:
The purpose of our study is to evaluate the effect of tramadol as an adjunct to ropivacaine local anesthetic solution in interscalene brachial plexus block for shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder surgery

Exclusion Criteria:

* patients on opioids
* diabetes mellitus
* interscalene block contraindicated
* patient refusing regional anesthesia techniques

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | 24 hours postoperatively

SECONDARY OUTCOMES:
Persistent postoperative pain | 1 month postoperatively, 3 months postoperatively
Evidence of motor blockade resolution, confirmed by elbow - wrist - fingers active movement | 24 hours postoperatively
Evidence of sensory blockade resolution, confirmed by pin-prick test | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepieion Hospital of Voula, Athens, Attica, Greece

REFERENCES:
- [Background] Lin E, Choi J, Hadzic A. Peripheral nerve blocks for outpatient surgery: evidence-based indications. Curr Opin Anaesthesiol. 2013 Aug;26(4):467-74. doi: 10.1097/ACO.0b013e328362baa4. PMID 23820103
- [Background] Bishop JY, Sprague M, Gelber J, Krol M, Rosenblatt MA, Gladstone JN, Flatow EL. Interscalene regional anesthesia for arthroscopic shoulder surgery: a safe and effective technique. J Shoulder Elbow Surg. 2006 Sep-Oct;15(5):567-70. doi: 10.1016/j.jse.2006.01.009. PMID 16979050